CLINICAL TRIAL: NCT00731081
Title: Observational Study About the Evolution of Severe Late Onset Pompe Disease Patient With Pulmonary Dysfunction and Receiving Myozyme
Brief Title: Study About the Evolution of Severe Late Onset Pompe Disease Patient With Pulmonary Dysfunction and Receiving Myozyme®
Status: Completed | Type: Observational
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: AGLU04107
Record Dates: First submitted 2008-08-06; First posted 2008-08-08 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-02

CONDITIONS: Pompe Disease (Late-Onset); Glycogen Storage Disease Type II (GSD II); Glycogenesis 2 Acid Maltase Deficiency
MeSH Terms: conditions — Glycogen Storage Disease Type II

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine and plasma oligosaccharides
Oversight: Data Monitoring Committee: No

SUMMARY:
To describe severe late onset patients with pompe disease receiving Myozyme®

ELIGIBILITY:
Inclusion Criteria:

* Male or Female ≥ 18 years of age;
* The patient and/or patient's legal representative has given their informed consent in writing before any study procedure is initiated;
* Pompe disease confirmed by documented deficit in endogenous acid alpha-glucosidase (GAA) activity;
* A severe form of the disease as defined as follows: a. Moderate to severe limb girdle muscle weakness requiring help for walking around (sticks, crutches, walking frame or wheelchair); and b. Symptoms of diaphragmatic dysfunction defined by at least 2 out of the 3 following criteria: orthopnea, vital capacity < 50%, paradoxical respiration detected in measurement of transdiaphragmatic pressure; and c. Use of invasive ventilation (defined by need for tracheotomy) or noninvasive ventilation (defined by utilization of assisted ventilation using a nasal or facial mask)day and night prescribed ≥ 12 hours/day;
* Treated for ≥6 months with Myozyme;
* Followed-up in a reference center according to the CETP recommendations.

Exclusion Criteria:

* The patient presents with a major congenital anomaly;
* The patient presents with a clinically important organic disease (except for symptoms related to Pompe disease) such as cardiovascular, hepatic, pulmonary, neurological or renal disease or any other medical condition, serious disease or particular circumstances that in the investigator's opinion, should preclude the patient's participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe late onset of Pompe disease with respiratory deficiency and treated by Myozyme
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2007-03; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
To describe severe late onset patients with Pompe disease receiving Myozyme and follow-up according to the CETP recommendations | 12 to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (1):
- Pitie-Salpetriere Hospital, Paris, France